CLINICAL TRIAL: NCT02729610
Title: The Use of Bronchial Blocker Versus Double Lumen Tube for One-lung Ventilation During Thoracoscope Assisted Mitral Valve Replacement
Brief Title: Bronchial Blocker for One-lung Ventilation in Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, HailongDong, Professor & Chief of Department of Anesthesiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20153001-1
Record Dates: First submitted 2016-03-21; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Complication of Ventilation Therapy; Intubation Complication; Postoperative; Dysfunction Following Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DLT group (Active Comparator): In this arm, patient will be intubated with a double lumen endotracheal tube
  Interventions: Device: double-lumen endotracheal tube (DLT group)
- BB group (Experimental): In this arm, patient will be intubated with an endobronchial blocker
  Interventions: Device: endobronchial blocker (BB group)

INTERVENTIONS:
Device: double-lumen endotracheal tube (DLT group) — In this arm, after anesthesia induction, a double lumen endotracheal tube will be intubated for one-lung ventilation
  Arms: DLT group
Device: endobronchial blocker (BB group) — In this arm, after anesthesia induction, an endobronchial blocker will be intubated for one-lung ventilation
  Arms: BB group

SUMMARY:
To investigate if bronchial blocker is more suitable for one-lung ventilation during thoracoscope assisted mitral valve replacement surgery with Cardiopulmonary Bypass than the double-lumen endobronchial tube.

DETAILED DESCRIPTION:
Postoperative hoarseness, sore throat, and vocal cord injuries are common complications after general anesthesia. The incidence of postoperative hoarseness is as frequent as 50% after short-term tracheal intubation. In the past, several risk factors for postoperative hoarseness and laryngeal injury have been identified, including demographic factors, quality of tracheal intubation and technical factors such as endotracheal tube size. One-lung ventilation during thoracotomy can be achieved via two basic techniques: (1) use of a double-lumen endotracheal tube (DLT) consisting of an endotracheal and an endobronchial lumen allowing independent single-lung ventilation ; or (2) use of an endobronchial blocker such as the Arndt blocker, which allows lung collapse distal to the occlusion. It has been recently demonstrated that DLT and endobronchial blocker are similar in their efficacy to achieve lung isolation for elective thoracic surgery. No data are available yet about the influence of the chosen technique on postoperative hoarseness, vocal cord injuries, sore throat, and bronchial injuries. Published data of Stout et al. imply that the incidence of postoperative hoarseness and vocal cord injury might be directly correlated with size of the used endotracheal tube. During thoracoscope assisted mitral valve replacement cardiac surgery, excellent lung isolated was not required. One-lung ventilation with the other lung collapsed is used to achieve a better exposure and assist the surgery. During the cardiac surgery under cardiopulmonary bypass, heparinization will lead to uncontrolled hemorrhage if there is endotracheal tube insertion associated injury. In addition, DLTs need to be exchanged for a single-lumen tube before the patient transferring to cardiac care unit for postoperative ventilatory support. This may result in second time injury. Investigators hypothesized that using a bronchial blocker to achieve one-lung ventilation may result in a lower incidence of clinically relevant laryngeal and bronchial morbidity after thoracoscope assisted mitral valve replacement cardiac surgery compared with a control group intubated with a DLT.

ELIGIBILITY:
Inclusion Criteria:

1. New York Heart Association (NYHA)I-III level.
2. scheduled for thoracoscope assisted mitral valve surgery under surgery
3. provide with informed consent.

Exclusion Criteria:

1. emergency surgery.
2. preoperative pulmonary diseases, such as chronic obstructive pulmonary disease, atelectasis.
3. preoperative voice hoarse or sore throat.
4. involved in other clinical trials within 3 months .
5. Cannot cooperate with language understanding disorders or psychological problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
clinically relevant laryngeal and bronchial morbidity | perioperative period
  incidence of clinically relevant laryngeal and bronchial morbidity will be recorded, including postoperative hoarseness, sore throat, and vocal cord injuries, pulmonary complications

SECONDARY OUTCOMES:
Heart Rate | perioperative period
  Heart rate in BPM will be recorded at right before intubation (T1), at intubation (T2), and at three minutes after intubation (T3).
Central Venous Pressure | perioperative period
  Central venous pressure in cmH2O will be recorded at right before intubation (T1),at intubation (T2), and at three minutes after intubation (T3).
Blood Pressure | perioperative period
  Systolic blood pressure, diastolic blood pressure and mean arterial pressure all in mmHg will be recorded at right before intubation (T1),at intubation (T2), and at three minutes after intubation (T3).
the Duration of Ventilation | The duration of ventilation in minutes will be recorded at time from intubation to extubation, an expected average of 18 hours.
  It is the duration of ventilation, prolonged ventilation is defined as patients remaining on the ventilator for more than 48 hours
Length of Postoperative Hospital Stay | Length of postoperative hospital stay in days will be recorded which is defined as the time from surgery to hospital discharge, an expected average of 10 days
  Recorded the time of postoperative hospital stay in days.
Length of CCU Stay | Length of CCU stay in hours will be recorded which is defined as the time stay in the cardiac intensive care unit, an expected average of 3 days.
  It is the length of stay in cardiac ICU

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD & PhD, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoo JY, Kim DH, Choi H, Kim K, Chae YJ, Park SY. Disconnection technique with a bronchial blocker for improving lung deflation: a comparison with a double-lumen tube and bronchial blocker without disconnection. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):904-7. doi: 10.1053/j.jvca.2013.07.019. Epub 2013 Nov 11. PMID 24231197
- [Background] Kuo AS, Philip JH, Edrich T. Airway ventilation pressures during bronchoscopy, bronchial blocker, and double-lumen endotracheal tube use: an in vitro study. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):873-9. doi: 10.1053/j.jvca.2013.03.023. Epub 2013 Sep 7. PMID 24021918
- [Background] Guo C, Ma C, Yu L. [Comparative of coopdech bronchial blocker and double-lumen tube on one lung ventilation in children]. Zhonghua Yi Xue Za Zhi. 2014 Jun 3;94(21):1651-3. Chinese. PMID 25152290
- [Background] Rothfield KP, Russo SG. Videolaryngoscopy: should it replace direct laryngoscopy? a pro-con debate. J Clin Anesth. 2012 Nov;24(7):593-7. doi: 10.1016/j.jclinane.2012.04.005. PMID 23101777
- [Background] Ruetzler K, Grubhofer G, Schmid W, Papp D, Nabecker S, Hutschala D, Lang G, Hager H. Randomized clinical trial comparing double-lumen tube and EZ-Blocker for single-lung ventilation. Br J Anaesth. 2011 Jun;106(6):896-902. doi: 10.1093/bja/aer086. Epub 2011 Apr 14. PMID 21493621
- [Background] Lei Q, Zeng QS, Zhang XS, Xie B, Luo ZC, Guo HM, Chen JM, Zhuang J. Superior vena cava drainage during thoracoscopic cardiac surgery: bilateral internal jugular vein sheaths versus one percutaneous superior vena cava cannula. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):914-8. doi: 10.1053/j.jvca.2013.05.043. Epub 2013 Oct 16. PMID 24139456